CLINICAL TRIAL: NCT01323842
Title: Hydro II: Emergency Department Ultrasound in Renal Colic
Brief Title: Emergency Department Ultrasound in Renal Colic
Status: Completed | Type: Observational
Sponsor: Queen's University (Other)
Collaborators: Ontario Ministry of Health and Long Term Care (Other Government)
Responsible Party: Principal Investigator, Dr. Marco L.A. Sivilotti, Research Director, Queen's University
Other Study IDs: Hydro II
Record Dates: First submitted 2011-03-24; First posted 2011-03-28 (Estimated); Last update posted 2015-11-26 (Estimated); Status verified 2015-11

CONDITIONS: Renal Colic; Hydronephrosis; Abdominal Aortic Aneurysm
Keywords: renal colic; hydronephrosis; abdominal aortic aneurysm; ultrasound; emergency medicine; urolithiasis
MeSH Terms: conditions — Renal Colic; Hydronephrosis; Aortic Aneurysm, Abdominal; Urolithiasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- rule in renal colic: ED patients with abdominal/flank pain where a diagnosis of renal colic is being considered and undergoing formal imaging while in the ED
  Interventions: Procedure: EDTU

INTERVENTIONS:
Procedure: EDTU — bedside ultrasound imaging by the treating emergency physician

SUMMARY:
Renal colic is a common (1300 visits per year at our institution) and painful condition caused by stones in the kidney and ureter, and can be mimicked by life threatening conditions such as a ruptured abdominal aortic aneurysm (AAA). This can create clinical uncertainty. Emergency department targeted ultrasound (EDTU) is performed by an emergency physician at the patient's bedside, and has been shown to be accurate, safe, and efficient. We have shown that EDTU can accurately identify hydronephrosis, which is a predictor of complications of kidney stones. A normal formal ultrasound (US) predicts an uncomplicated clinical course. We will assess the accuracy of EDTU for the diagnosis of hydronephrosis, and when normal, whether patients can be safely discharged.

ELIGIBILITY:
Inclusion Criteria:

* Age 16 - 65 years
* Symptoms suggestive of renal colic
* EDTU performed within one hour (before or after) of formal imaging
* Imaging study arranged during this ED visit (includes next morning)

Exclusion Criteria:

* Hemodynamic instability (Pulse > 120 or SBP < 90 or requiring vasopressors)
* Fever (>38 degrees C)
* Leukocytes and nitrites on dipstick urinalysis (evidence of urinary tract infection)
* Pregnancy
* Inmate
* Renal transplant or single functioning kidney

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: ED patients with suspected renal colic being imaged while in the ED
Sampling Method: Non-Probability Sample
Enrollment: 414 (Actual)
Dates: Start 2011-03; Primary Completion 2013-07 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
complications post-ED visit in patients with and without negative EDTU. | 30 days
  The frequency of complications by 30 days post-ED visit in patients with and without negative EDTU.
diagnostic accuracy for hydronephrosis | 1 hours
  The accuracy of ED physicians in using EDTU to assess for hydronephrosis when compared to diagnostic imaging by CT or formal ultrasound.

SECONDARY OUTCOMES:
ED length of stay | 1 day
  estimates of potential time of ED stay saved if a clinical decision is made on the basis of an EDTU (rather than waiting for formal diagnostic imaging)
radiation dose | 1 hour
  potential savings in radiation exposure from avoiding CT scanning
accuracy in ruling out AAA | 1 hour
  accuracy of ED physicians in using EDTU to assess aortic size (and rule out AAA) when compared to diagnostic imaging by CT or formal ultrasound will also be validated.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Bruder, MD, Principal Investigator — Queen's University
Locations (1):
- Kingston General Hospital, Kingston, Ontario, Canada

REFERENCES:
- [Derived] Sibley S, Roth N, Scott C, Rang L, White H, Sivilotti MLA, Bruder E. Point-of-care ultrasound for the detection of hydronephrosis in emergency department patients with suspected renal colic. Ultrasound J. 2020 Jun 8;12(1):31. doi: 10.1186/s13089-020-00178-3. PMID 32507905